CLINICAL TRIAL: NCT03350100
Title: An Investigation Into the Acute Effects of Date Fruit (Phoenix Dactylifera L.) on Mood and Cognitive Performance in Healthy Volunteers.
Brief Title: The Effect of Date Fruit on Mood and Cognition in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DFCPM1
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Mood and Cognitive Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Birhi date cultivar (Experimental): A 48.46 g of freeze dried powder of Birhi date Cultivar which is equivalent to a 115g of fresh dates, contains 14.72 g of total sugar in which 4.6 g Glucose, 2.49 fructose and 3.4 sucrose, and a total phenolic content of 162.8 mg/100 g of GAE. and 0.80 g of fibres, will be mixed into one portion of low fat yogurt (e.g. Yeo yogurt 150 g BigFish®, which gives a total energy of 299 KJ.
  Interventions: Dietary Supplement: Acute effect of two Saudi cultivars of date fruit on mood and cognitive performance
- Khassab date cultivar (Experimental): A 34.5 g of freeze dried powder of Khassab date Cultivar which is equivalent to A 115g of fresh dates, contains 14.72 g of total sugar in which 4.6 g Glucose, 2.49 fructose and 3.4 sucrose, and a total phenolic content of 91.52 mg/100 g of GAE. and 0.80 g of fibres,will be mixed into one portion of low fat yogurt (e.g. Yeo yogurt 150 g BigFish®, which gives a total energy of 299 KJ.
  Interventions: Dietary Supplement: Acute effect of two Saudi cultivars of date fruit on mood and cognitive performance
- placebo (Placebo Comparator): A 14.72 g of total sugar in which 4.6 g Glucose, 2.49 fructose and 3.4 sucrose, and 0.80 g of fibres, will be mixed into one portion of low fat yogurt (e.g. Yeo yogurt 150 g BigFish®, which gives a total energy of 299 KJ.
  Interventions: Dietary Supplement: Acute effect of two Saudi cultivars of date fruit on mood and cognitive performance

INTERVENTIONS:
Dietary Supplement: Acute effect of two Saudi cultivars of date fruit on mood and cognitive performance — Acute effect of two Saudi cultivars of date fruit on mood and cognitive performance at baseline, 45 post-dose, 90 min post-dose and 135 min post-dose

SUMMARY:
A number of studies have considered the neuroprotective effects of date fruit on neurodegenerative diseases in animals. However, so far no study has addressed the acute effects of date fruit on mood and cognitive performance in humans. This study will investigate the acute effects of two different cultivars of Saudi dates on mood and cognitive performance into healthy volunteers.

This study will follow a double blind, randomised, placebo controlled, repeated measures, cross over design with two active treatment arms versus placebo. Treatment orders will be counterbalanced with the use of a Latin Square design.

Thirty six healthy participants aged between 18 and 35 will be recruited. Participants will be required to undergo a screening/training visit, followed by three measurement visits at weekly intervals. The trial will last for 3 months in total.

DETAILED DESCRIPTION:
Introduction Fruit of the date palm (P. dactylifera) may be considered an emerging and potential candidate for the development of health-promoting foods owing to its high nutritive values (Juhaimi, Ghafoor et al. 2012). Recently, scientific studies have revealed the medicinal properties of P. dactylifera in the different ripening stages by examining anti-inflammatory, anti-angiogenic and antibacterial activity. The anti-inflammatory activity of various parts of P. dactylifera have been evaluated (Shabani, Zangiabadi et al. 2013); it is evident from these studies that, both in vivo and in vitro, date fruits display anti-inflammatory activity, strongly linked to secondary metabolites and antioxidant behaviour.

More than 16 published studies have investigated the physiological and the psychological effects of P. dactylifera on the brain using animal models. Although this domain of research is in its infancy , the findings are quite promising and suggest that date fruits have the potential to become, on the one hand, a neuroprotective agent in ischemic stroke (Majid, Marzieh et al. 2008), brain damage (Kalantaripour, Asadi-Shekaari et al. 2012), and Alzheimer's disease and (Essa, Akbar et al. 2016), on the other hand, a brain enhancer by attenuating impairment in cognition caused by neurodegenerative diseases (Subash, Essa et al. 2015).

Aim The aim of this study is to investigate the acute effects of two different cultivars of P. dactylifera commonly consumed in Saudi Arabia on mood and cognitive performance of healthy volunteers.

Design The project will investigate the acute effects on human cognitive function and mood after the administration of a single dose of two different date fruits using a yogurt as the carrier medium against a control yoghurt matched for sugar, flavour, volume, fibers, taste and appearance. The study will follow a double-blind, counterbalanced, placebo controlled, repeated measures design, with two active treatment arms versus placebo, with one week between each measurement visit. Treatment orders will be counterbalanced with the use of a Latin Square design (Williams 1949). Participants will be randomly allocated to a treatment order as selected through a Williams Latin Square. Participants will be required to undergo a screening/training visit, followed by three measurement visits at weekly intervals. The trial will last for 3 months in total, which is about 2-3 weeks for each participants.

Treatment Five different cultivars of date fruit were initially considered and screened for testing against cognitive performance and mood according to the following criteria; popularity, representation of the different maturation stages, and representation of the different colours, which has a great an effect on the total phenolic content. Therefore from the Bisir maturation stage Khasab and Birhi dates were chosen, from the Rutab maturation stage Sukari dates and Ajwah and Khalas dates were chosen from the Tamer maturation stage.

After a chemical analysis of polyphenol content of the five different cultivars, the study was narrowed down to two different cultivars of date fruits: Khasab and Birhi. According to our initial analysis Khasb and Birhi cultivars contained the highest amount of polyphenols, and while the total sugar in all varieties was similar it was lower in these two varieties compared with the others tested.

Taking the stickiness of the fruit and the high content of fibres, a total of 115g of date powder will be mixed into one portion of low fat yogurt (e.g. Yeo yogurt 150 g BigFish® which has 240kJ/56kcal), with consideration to the wet weight variation prior to freeze drying process. The naturally occurring sugars in the date will be quantified. The total volume of the treatment yogurt will be up to 265 mg. The control yogurt will be a placebo mix containing glucose, fructose, sucrose, fibres and food dye in order to be closely matched for volume, taste, appearance, texture, and energy with the treatment. Yogurts will be coded and prepared freshly each morning by a third party who shall not take further part in the running of the study. No member of the investigation team will be aware of the coding of the drinks until a blind-data review is completed. Both the treatments and the placebo will be provided to the participants in plastic cups of similar appearance.

Participants A total of 36 healthy participants aged between 18 and 35 will be recruited through advertisement via poster and flyer. All participants will be required to undergo a screening visit.

Study procedures:

1. Screening All participants will be screened for any contraindications prior to the beginning of the study. The eligible participants will then be asked to complete the Cog-Track Battery four times to remove practice effects. On each of the study days, cognitive assessments will be conducted at baseline, 45 min post dose, 90 min post dose and 135 min post dose. After completing each cognitive assessment, participants will be asked to complete Visual Analogue Scales to assess their mood status.
2. Study day The volunteers will be briefed about the study protocol and will sign a written informed consent (see appendix). The participants will arrive at the NU-Food research center at about 9:30 am after a 12 hour overnight fast. Measurements of height and weight will be taken again in order to track any change, and this will be followed by a completion of the baseline Cog-Track Battery, Bond-Lader Visual Analogue Scales, Profile of mood states questionnaire and finger-prick blood glucose test. The participants will then consume their treatment for that day (as allocated by the Williams Latin square) and be asked to sit quietly (participants may work quietly, read or watch TV as they wish). They will be asked to start the second period of cognitive performance tasks 45 min after treatment administration to coincide with another blood glucose test. The same tasks (cognition and blood glucose) will be collected again at 90 min and 135 min post dose. Each of the three study visits will last approximately 3 hours. Participants will be required to stay in the research center during breaks between each test/blood sample. Participants will have access to a comfortable waiting room. At the end of the testing day all participants will receive a standard meal (A sandwich and a drink). (A detailed scheduling for screening and study days can be found in appendixes).

ELIGIBILITY:
Inclusion Criteria:

A total of 36 healthy participants aged between 18 and 35 will be recruited through advertisement via poster and flyer. All participants will be required to undergo a screening visit.

Exclusion Criteria:

Healthy participants aged 18-35 with a BMI >18 <36 will be recruited from the Newcastle Upon-Tyne area

Participants will be considered ineligible to participate in the study if they meet any of the following criteria:

1. They have a BMI above 35kg/m2 or lower than 18kg/m2
2. They smoke or consume tobacco products
3. They are taking any illicit or prescribed drugs
4. They are using dietary supplements, over the counter medicine or recreational drugs
5. They have a history of or currently abuse alcohol
6. They have a history of dyslexia, ADHD, learning difficulties or color blindness
7. They are females who are pregnant, seeking to become pregnant or do not use
8. They have allergies to any food products.
9. They have any metabolic diseases such as type 1 or type 2 diabetes.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
cognition: Simple Reaction Time | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Cog-track an online set of nine cognitive tests (www.wesnes.com).
Cognition: Digit Vigilance | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Cog-track an online set of nine cognitive tests (www.wesnes.com).
Cognition: Choice Reaction Time | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Cog-track an online set of nine cognitive tests (www.wesnes.com).
Cognition: Numeric Working Memory | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Cog-track an online set of nine cognitive tests (www.wesnes.com).
Cognition: Spatial Working Memory | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Cog-track an online set of nine cognitive tests (www.wesnes.com).
Cognition: Immediate Word Recall | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Cog-track an online set of nine cognitive tests (www.wesnes.com).
Cognition:Delayed Word Recall | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Cog-track an online set of nine cognitive tests (www.wesnes.com).
Cognition:Word Recognition | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Cog-track an online set of nine cognitive tests (www.wesnes.com).
Cognition:Pattern Separation | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Cog-track an online set of nine cognitive tests (www.wesnes.com).
Mood scales Bond Lader | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  The Bond and Lader Visual Analogue Scales (1974)
The Profile of Mood States (POMS) | Change from visit 1 to visit 2 to visit 3
  The Profile of Mood States (POMS; McNair et al., 1992)
Blood Glucose level test | Change from baseline, 45 min pos-dose, 90 min post-dose and 135 postdose
  Finger prick

CONTACTS AND LOCATIONS:
Locations (1):
- NU-Food Research Facility, Newcastle upon Tyne, Tyne and Wear, United Kingdom